CLINICAL TRIAL: NCT02680535
Title: A Study of MRI/US Fusion Imaging and Biopsy in Combination With Nanoparticle Directed Focal Therapy for Ablation of Prostate Tissue
Brief Title: MRI/US Fusion Imaging and Biopsy in Combination With Nanoparticle Directed Focal Therapy for Ablation of Prostate Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanospectra Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-PC-002
Record Dates: First submitted 2016-02-02; First posted 2016-02-11 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Neoplasms of the Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AuroShell particle infusion (Experimental): Single intravenous infusion of AuroShell particles 12 to 36 hours prior to ultrasound-guided laser irradiation using a FDA cleared laser and an interstitial optical fiber.
  Interventions: Device: AuroShell particle infusion

INTERVENTIONS:
Device: AuroShell particle infusion — Infuse AuroShell particles for irradiation by AuroLase laser to ablate neoplasms of the prostate.

SUMMARY:
To determine the efficacy of using MRI/US fusion imaging technology to direct focal ablation of prostate tissue using nanoparticle-directed laser irradiation.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single-dose study of AuroLase Therapy in the focal ablation of neoplastic prostate tissue via nanoparticle directed irradiation. The patient population consists of men with low to intermediate risk localized prostate cancer with MRI visible and confirmed focal areas of prostate cancer using MR US Fusion Guided Biopsy. The patient also has no disease detected via ultrasound guided biopsy outside of areas visualized on MR imaging.There is one arm/group to this study: Up to forty five (45) patients will receive a single intravenous infusion of AuroShell particles 12 to 36 hours prior to MRI/US guided laser irradiation using an FDA cleared laser and an interstitial optical fiber.

Efficacy and acute volume of ablation will be assessed by contrast-enhanced MRI 48 - 96 hours after laser illumination to allow time for the appearance of coagulative necrosis and prior to reconfiguration of tissue by lytic action. An appearance of a 'void' on MRI would be more generally expected than lesion shrinkage. Efficacy of focal ablation of prostate tissue will be assessed by MRI /Ultrasound guided biopsy at 3 months (primary endpoint) and again at 1 year after laser treatment. Per standard of care patient follow up will continue on a 6 month basis beyond the one year follow up but will be outside the scope of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented histological or cytological evidence of tumor(s) of the prostate.
* Patients must be ≥ 45 years of age
* Patients or their legal representative must be able to read, understand and sign an informed consent
* Organ confined clinical T1C or clinical T2a prostate cancer that is visualized on MR imaging
* Prostate cancer is diagnosed by MR image guided biopsies
* Gleason Score ≤ 7; and 2 or less positive lesions on prior MR US fusion guided prostate biopsy.
* If the standard biopsy cores are positive, they must be from the same location in the prostate as MR lesion was biopsied and proven to be cancerous. (Left / Right, Base, Mid Gland, Apex).
* Prior MRI results dated within 120 days prior to ablation.
* No metastatic disease as per NCCN guidelines (www.nccn.org) - Bone scan indicated to r/o metastatic disease if clinical T1 and PSA > 20 or T2 and PSA > 10
* PSA < 15 ng/ml or PSA density < 0.15 ng/ml2 in patients with a PSA > 15 ng/ml
* The patient has given written informed consent after the nature of the study and alternative treatment options have been explained

Exclusion Criteria:

* Patients with known hypersensitivity to any of the components of the PEGylated AuroShell suspension (polyethylene glycol, gold)
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within a period of 5 half-lives of the investigational therapy in question prior to the day of dosing with the PEGylated AuroShell particles (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Patients with evidence of an active bacterial infection or with a fever ≥ 38.5 ºC (101.3 ºF) within 3 days of the first scheduled day of dosing
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* The presence of 3 or more MR Visible lesions positive on biopsy.
* The presence of extra capsular, seminal vesicle invasion or metastatic disease.
* Patient is unable to tolerate MRI (foreign body; i.e. pacemaker or other implanted device; claustrophobia; inability to tolerate rectal coil, etc…)
* Patient with inability to follow up.
* History of prior treatment for prostate cancer.
* Acute urinary tract infection.
* Lower urinary tract symptoms defined by International Prostate symptom score (IPSS) > 20
* Patients with renal insufficiency with an estimated glomerular filtration (EGF) <= 30 are excluded, due to they will not be able to undergo gadolinium enhance MRI.
* Patients with acute or chronic hepatic dysfunction as evidenced by clinically significant abnormalities in albumin, total protein, or prothrombin time, or evidence of hepatic injury with clinically important (> grade 1) changes in AST, ALT, ALP, bilirubin, or GGT values.
* Patients with uncontrolled coagulopathies who are at increased risk of bleeding.
* Altered mental status preventing consent or answering questions during conduct of the trial will be excluded for safety purposes.
* Other medical or surgical conditions, especially involving the cardiac, respiratory, renal or hepatic organ systems that would either be unsafe for the patient, would limit study participation, or that would impede the determination of causality of any adverse events experienced during the conduct of this study.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Evidence of efficacy of focal ablation of clinically significant targeted prostate lesion(s) confirmed using 3T MRI/Ultrasound guided biopsy 3 months after treatment. | Three Months
  Efficacy of focal ablation will be assessed by 3T MRI/Ultrasound guided biopsy at 3 months after treatment. Focal ablation of clinically significant targeted prostate lesions(s) as confirmed with negative biopsies with minimal damage to surrounding healthy tissue.

SECONDARY OUTCOMES:
Adverse Events | Start to Three Months
  Any adverse device effects attributable to near infrared illumination of the prostate following AuroShell particle infusion.
Evidence of efficacy of focal ablation of clinically significant targeted prostate lesion(s) confirmed using 3T MRI/Ultrasound guided biopsy one year after treatment. | One Year
  Efficacy of focal ablation will be assessed by 3T MRI/Ultrasound guided biopsy at one year after treatment. Focal ablation of clinically significant targeted prostate lesions(s) as confirmed with negative biopsies with minimal damage to surrounding healthy tissue.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of Texas Medical Branch, Galveston, Texas
  - University of Texas Medical School at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jue JS, Coons S, Hautvast G, Thompson SF, Geraats J, Richstone L, Schwartz MJ, Rastinehad AR. Novel Automated Three-Dimensional Surgical Planning Tool and Magnetic Resonance Imaging/Ultrasound Fusion Technology to Perform Nanoparticle Ablation and Cryoablation of the Prostate for Focal Therapy. J Endourol. 2022 Mar;36(3):369-372. doi: 10.1089/end.2021.0266. Epub 2021 Sep 13. PMID 34409850